CLINICAL TRIAL: NCT01773772
Title: Progesterone Suppression of Nocturnal LH Increases in Pubertal Girls (JCM017)
Brief Title: Progesterone Suppression of Nocturnal LH Increases in Pubertal Girls
Acronym: JCM017
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chris McCartney, Associate Professor, Department of Medicine, Endocrinology and Metabolism, University of Virginia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 10504; U54HD028934 (NIH); P50HD028934 (NIH)
Record Dates: First submitted 2012-05-17; First posted 2013-01-23 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Female Puberty
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Progesterone (Experimental): Subjects will take 25-50 mg oral micronized P or placebo at 1600 h and again at 2000 h. P dosing will be based on weight, with 25 mg administered to girls < 42kg and 50 mg given to those > or = 42 kg.
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): Subjects will take placebo at 1600 h and again at 2000 h.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — Subjects will take 25-50 mg oral micronized progesterone at 1600 h and again at 2000 h. Progesterone dosing will be based on weight, with 25 mg administered to girls < 42kg and 50 mg given to those or = to 42 kg.
  Arms: Progesterone
Drug: Placebo — Subjects will take oral placebo suspension at 1600 h and again at 2000 h.
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn more about how gonadotropin-releasing hormone (GnRH) and luteinizing hormone (LH) pulses are controlled during puberty. In this study, the investigators aim to discover whether or not giving 2 small doses of progesterone to early pubertal girls will prevent the nighttime increase of GnRH and LH pulses. From the information gathered in this study, the investigators may be able to learn more about how menstrual cycles are normally established in girls during puberty. Ultimately, if these normal processes can be understood, the investigators may be able to better understand abnormalities of puberty.

DETAILED DESCRIPTION:
We will recruit early pubertal, premenarcheal adolescent girls, since these stages are associated with the most prominent diurnal variations in LH pulsatility (13). Weight will be normal for height (i.e., BMI ≤ 85th and ≥ 5th percentile for age according to the CDC), and plasma testosterone will be < 40 ng/dl. We will recruit normal adolescent girls, or girls with idiopathic short stature (> 2 SD below mean height for age with no identifiable cause), from UVa Pediatric Clinics, local pediatric clinics, the Teen Health Center, and UVa Endocrine Clinics. Subjects will be late Tanner 1 (defined as having estradiol level > 20 pg/mL), Tanner 2, or Tanner 3. All potential subjects will undergo a screening history and physical prior to enrollment. These 60-90 min outpatient visits to the CRU or alternate UVA clinical unit will establish general health and developmental normality. Evaluation will include a complete personal and family medical history and physical examination (including height, weight, and pubertal stage determination using the Tanner scale). The goals and procedures of the study will be explained to potential subjects and their parents, and questions will be entertained. The volunteer and her parents will sign the assent and consent forms, respectively. Blood (20 ml) will then be drawn (at approx. 0800-0900 h) for the following tests: LH, FSH, P, E2, total testosterone, SHBG, DHEA-S, 17-OHP, beta-hCG, TSH, CBC, chemistry and liver panels, prolactin, insulin, Insulin-like Growth Factor 1 (IGF-1), and cytokines and adipokines (including adiponectin, leptin, resistin, PAI-1, IL-1b, IL-6, IL-8, TNFa, MCP-1, HGF and NGF). Subjects will need to fast for a minimum of 8 hours prior to screening blood draw. Bone age (plain x-ray of left hand and wrist) will also be performed as a marker of biological age, since pubertal stage generally correlates better with bone age than chronological age.

If the screening labs show a hemoglobin < 11.0g/dL for African American subjects or hemoglobin < 11.5 g/dL for non-African American subjects, iron therapy at a dose of 1-2 mg/kg will be encouraged for 60 days. Subjects weighing ≤ 36 kg will be given 300-325 mg oral ferrous gluconate daily (containing 36 mg of elemental iron); subjects weighing > 36 kg will be given 300-325 mg oral ferrous gluconate twice daily. Hemoglobin will then be rechecked in the CRU or clinical unit; if acceptable (hemoglobin ≥ 11 g/dL for African American subjects or hemoglobin ≥ 11.5 g/dL for non-African American subjects), the inpatient admission will be scheduled.

If the screening labs are normal, iron supplementation at a dose of 1-2 mg/kg for 30 days will be given to help prevent anemia from developing during the study. Subjects weighing ≤ 36 kg will be given 300-325 mg oral ferrous gluconate daily (containing 36 mg of elemental iron); subjects weighing > 36 kg will be given 300-325 mg oral ferrous gluconate twice daily.

If safety labs are abnormal during screening (e.g., abnormal liver tests, abnormal TSH), subjects will be asked to return once for repeat (confirmatory) labs to exclude lab error. Repeat testing will generally occur within one month of the original screening lab draw. If exclusionary lab values are confirmed on such repeat testing, subjects will be excluded from participation.

1-3 days before overnight admission: An outpatient blood sample will be obtained 1-3 d before overnight admission. Plasma P will be checked to exclude an unlikely luteal phase, with overnight admission cancelled if P exceeds 1.5 ng/ml. Hemoglobin will be obtained if these have not been obtained within 30 days of the overnight admission (subsequent overnight admission cancelled if hemoglobin < 11 g/dl for African American subjects or < 11.5 g/dL for non-African American subjects). Urine beta-HCG will be assessed to exclude pregnancy. If three months have elapsed between an overnight admission and the subject's most recent safety labs, then additional safety labs (chemistry and liver panel) will be obtained at this time.

Inpatient Admission: Subjects will be admitted to the CRU, alternate UVA hospital unit, or off-site hotel at 1400 h. In general, parents are welcome to stay with their child at the off-site hotel if they wish. If the overnight portion of the study is to be done at an off-site hotel, the subject may stay without a parent or legal guardian, as long as two CRU staff are present. Whether or not a parent needs to remain during the overnight admission will be discussed when the visit is scheduled. An i.v. line with be placed in the forearm vein (this may be facilitated by EMLA cream), on the same side as the dominant hand if possible. Subjects will take 25-50 mg oral micronized P or placebo at 1600 h and again at 2000 h. P dosing will be based on weight, with 25 mg administered to girls < 42 kg and 50 mg given to those ≥ 42 kg; with P administration, we aim to produce mean P concentrations of approximately 2-3 ng/ml. Frequent blood sampling will begin at 1900 h and continue for 14 h as follows: LH every 10 min (1 ml); and FSH every 10 min (no additional blood required); P, E2, T, DHEA and cortisol every 30 min (1 ml). An additional 0.3 cc sample will be drawn at 0700 to test for fasting glucose. Fasting insulin, SHBG, estrone, androstenedione, DHEA-S will be performed on pooled samples from 05:00-07:00.

Lights will be extinguished at 2200 h to facilitate sleep, which will be carefully recorded by trained observers. During blood sampling, activity (e.g. awake, sleeping) will be recorded by the nurse every 10 minutes. Additionally, periods of sleep will be estimated using wrist actigraphy (Motionlogger Basic-L; Ambulatory Monitoring, Inc.) The Motionlogger Basic-L is a watch-like device (that includes an accelerometer) that will be worn on the non-dominant wrist by the research participant during the overnight admission. There will be an overnight fast from 22:00 until 07:00. Subjects will be awakened at 0700 h. Sampling will cease at 0900 h.

During the admission, ~150 ml of blood will be drawn (including 0.25 ml discarded with each sample). The total amount of blood that will be drawn during the study, including the screening, outpatient P sampling, and inpatient admission is ~170 ml. One of the parents will be allowed to stay overnight with the subject during the admission. After the last sample is taken, volunteers will be discharged on oral iron supplementation to be taken for 30 d.

Follow-up:

We will advance every effort to follow subjects (via outpatient CRU or clinic visits) at 6- to 12-month intervals for up to 3 y to assess progression of puberty, onset and frequency of menses, and development of signs of hyperandrogenism (e.g., hirsutism). We will obtain blood for LH, FSH, E2, P, and T during these follow-up visits. These follow-up visits will be encouraged, but not mandatory.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers in early to mid-puberty (i.e. late Tanner 1 [estradiol level >20 pg/ml], Tanner 2, or Tanner 3)
* Premenarcheal

Exclusion Criteria:

* BMI-for-age > 85th percentile or < 5th percentile
* Pregnancy
* Inability to comprehend what will be done during the study or why it will done
* Hyperandrogenism (e.g., hirsutism, elevated free testosterone level)
* History of allergy to progesterone (which is extremely rare)
* Hemoglobin less than 12 g/dl and hematocrit less than 36%
* Persistently abnormal sodium, potassium, or bicarbonate (i.e. confirmed on repeat)
* Persistently elevated creatinine, hepatic transaminases, or alkaline phosphatase (i.e., confirmed on repeat)
* Total bilirubin > 1.5 times upper limit of normal (i.e. confirmed on repeat)
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure; asthma requiring intermittent systemic corticosteroids; etc.)
* Untreated hypo- or hyperthyroidism, reflected by persistently abnormal thyroid-stimulating hormone (TSH) values
* Premature adrenarche (i.e., occurring before age 8 y)
* Basal (follicular) 17-hydroxyprogesterone > 200 ng/ml (confirmed on repeat)
* Dehydroepiandrosterone-sulfate (DHEA-S) > age-appropriate upper limit of normal (confirmed on repeat)
* Hyperprolactinemia (confirmed on repeat)
* Weight less than 25 kg

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2005-02-08 (Actual); Primary Completion 2009-06-08 (Actual); Study Completion 2009-06-08 (Actual)

PRIMARY OUTCOMES:
LH pulse frequency (number of LH pulses per hour) | 19 hours [from 1400 hr to 0900 hr]

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. McCartney, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Research in Reproduction, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No